CLINICAL TRIAL: NCT01327586
Title: Abstinence-Linked Money Management Multisite
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0904004971; R01DA012952 (NIH)
Record Dates: First submitted 2011-02-02; First posted 2011-04-01 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2014-07

CONDITIONS: Dual Diagnosis; Cocaine Abuse; Cocaine Dependence; Polysubstance Abuse
Keywords: disability; substance abuse; cocaine abuse; dual diagnosis; representative payee; HIV risk reduction
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATM (Experimental): Advisor-Teller Money Manager
  Interventions: Behavioral: ATM
- Individual Drug Counseling (Active Comparator)
  Interventions: Behavioral: Individual Drug Counseling

INTERVENTIONS:
Behavioral: ATM — Weekly counseling focused on improving money management, abstaining from cocaine,and minimizing unprotected sex
  Arms: ATM
Behavioral: Individual Drug Counseling — Standard individualized drug counseling, modified from that described by Woody and colleagues
  Arms: Individual Drug Counseling

SUMMARY:
Randomized clinical trial comparing a money management-based intervention involving storage and management of client funds, substance abuse counseling, and risk reduction counseling to individualized drug counseling.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in ambulatory psychiatric treatment at one of the participating clinics
* Receives SSI or SSDI payments
* Able to provide written informed consent
* Cocaine use within the last 60 days as evidenced by either a positive toxicology screen or self-reports

Exclusion Criteria:

* Has a conservator of person
* A history of violence towards clinical providers or predatory violence
* Suicidal plans or intent; homicidal plans or intent. Suicidal or homicidal ideation will not be exclusion criteria
* Physiological dependence on alcohol, illicit opiates or illicit sedatives as evidenced by a history of four weeks of daily use of these substances; and either tolerance or withdrawal (as defined by DSM IV-TR). The "standard withdrawal scales" referred to in DSM IV-TR will be the CIWA-AR (Sullivan et al., 1989) and the Clinical Opiate Withdrawal Scale (Wesson and Ling, 2003), with P.I. review because signs on the CIWA-AR such as "aware of sounds around you" may reflect psychiatric illness, not withdrawal
* Will not be able to complete the twelve months of the study because of anticipated incarceration or move
* Had been enrolled in the ongoing study
* Unable to speak and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2009-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Proportion of Urine toxicology tests without cocaine | Month 0,1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12

SECONDARY OUTCOMES:
Unprotected sexual encounters | Month 0, 1,2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  ACASI-measured

CONTACTS AND LOCATIONS:
Overall Officials: Marc I Rosen, M.D., Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Greater Bridgeport Mental Health Center, Bridgeport, Connecticut
  - Capitol Region Mental Health Center, Hartford, Connecticut